CLINICAL TRIAL: NCT01745445
Title: Phase ⅡClinical Trial of Randomized Concurrent Chemoradiotherapy or Radiotherapy Alone for Local-advanced Small Cell Lung Cancer After Induced Chemotherapy
Brief Title: Clinical Randomized Study of Concurrent Chemo-radiotherapy vs Radiotherapy Alone to Local-advanced Small Cell Lung Cancer (SCLC)
Acronym: SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIH-PQS-201205001
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-04

CONDITIONS: Small Cell Lung Cancer
Keywords: limited-stage small cell lung cancer; concurrent chemo-radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiotherapy alone arm (Experimental): VP-16 50 mg/m2 on day 1-5 and Carboplatin AUC = 5 on day 1 will be given by intravenous infusion for 3-4 cycles. Then a total dose of 60 Gy will be given in 30 fractions of 2 Gy, 5 fractions per week; All patients will be radiated by external beam radiation, using 3-D conformal radiation technique.
  Interventions: Other: concurrent chemo-radiotherapy arm

INTERVENTIONS:
Other: concurrent chemo-radiotherapy arm — VP-16 50 mg/m2 on day 1-5 and Carboplatin AUC = 5 on day 1 will be given by intravenous infusion for 3-4 cycles. Then a total dose of 60 Gy will be given in 30 fractions of 2 Gy, 5 fractions per week; Starting the first cycle of concurrent chemotherapy at the first day of radiotherapy. The chemotherapeutic scheme is intravenous infusion of Cisplatin 25mg/m2 on day 1-3 and oral administration of Etoposide 100mg on day1-5 and 3 weeks as a cycle for 2 consecutive cycles.

SUMMARY:
This trial aims to evaluate the efficacy and safety between radiotherapy alone and concurrent chemo-radiotherapy after 3-4 cycles of chemotherapy in LS-SCLC.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) represents 15-30% of all lung malignancies in China. Limited-stage small cell lung cancer (LS-SCLC) represents approximately 40% of cases. The current standard of care in limited-stage disease is systemic chemotherapy plus concurrent thoracic radiotherapy. Early concurrent chemo-radiotherapy is recommended for patients with limited-stage SCLC based on randomized trials. But, the administration of thoracic radiotherapy requires the assessment of several factors, including the volume of the radiation port, dose of radiation, and fractionation of radiotherapy. Parts of the LS-SCLC are local advanced stage (stage Ⅲa and Ⅲb), which can not tolerate concurrent chemo-radiotherapy because of large size in tumor and extensive metastasis of lymph nodes. At present, it is usually use 3-4 cycles of introduction chemotherapy to decrease the tumor size followed by definitive radiotherapy. But it is unclear whether this scheme is tolerant well or it could improve the overall survival in patients with LS-SCLC. As a result, we designed a prospective phase II randomized controlled trial in order to compare the tolerance and therapeutic effects between radiotherapy alone and concurrent chemo-radiotherapy after 3-4 cycles of chemotherapy in LS-SCLC.

ELIGIBILITY:
Inclusion Criteria:

Age 18- 75 years; ECOG performance status 0 or 1; Pathological or cytological confirmation of SCLC; Local stage small cell lung cancer with stage Ⅲa and Ⅲb; Receive 3-4 cycles of chemotherapy with etoposide plus cisplatin; Measurable disease using RECIST criteria with at least one lesion;

Adequate hematological, renal, hepatic and pulmonary functions defined as:

granulocytes ≥ 2.0×109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 8g/L, total bilirubin ≤ 1.5 x upper normal limit, aspartate aminotransferase, alanine aminotransferase≤2.5 × upper normal limit,, creatinine ≤ 1.5mg/L, FEV1 ≥ 1.5 L Ability to understand and willingness to sign a written informed consent form;

Exclusion Criteria:

History of operation of lung cancer; PD after 3-4 cycles chemotherapy; Patients with sever infection; Patients with uncontrollable diabetes; Patients in pregnancy or lactation; Patients who are currently receiving or have received other clinical trail for radioprotection within the prior six months are excluded; Patient with history of malignancy other than skin cancer or Carcinoma in-situ within 2 years; History of cardiovascular diseases that might include one of the following: myocardial infraction, angina, coronary angioplasty, congestive heart failure, stroke, or coronary bypass surgery in the last 6 months; Concomitant treatment with other anticancer drugs;

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years
  DFS was defined as the length of time from the date of randomization to the date of first documentation of relapse of SCLC or any other type of cancer or death.

SECONDARY OUTCOMES:
overall survival | 3 years
  OS was defined as the length of time from the date of randomization to the date of death of various reasons.
acute and late toxic effects | 3 months and 3 years
  acute toxic effect was defined as toxic effects less than 90 days from initiation of treatment late toxic effect was defined as toxic effects more than 90 days from initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: QING SONG PANG, M.D, Study Director — Department of Radiation Oncology, Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao J, Zhang W, Er P, Chen X, Guan Y, Qian D, Wang J, Yuan Z, Zhao L, Wang P, Pang Q. Concurrent or Sequential Chemoradiotherapy after 3-4 Cycles Induction Chemotherapy for LS-SCLC with Bulky Tumor. J Cancer. 2020 Jun 16;11(17):4957-4964. doi: 10.7150/jca.41136. eCollection 2020. PMID 32742443